CLINICAL TRIAL: NCT06583031
Title: A Phase 1, Randomized, Modified Double-blind, Multi-center, Parallel Group, Multi-arm Study to Investigate the Safety and Immunogenicity of an RSV/hMPV Vaccine Candidate in Adult Participants Aged 60 to 75 Years
Brief Title: Study to Evaluate the Safety and Immune Response of an Investigational Vaccine for the Prevention of RSV (Respiratory Syncytial Virus) and (hMPV) Human Metapneumovirus Infection in Participants Aged 60 to 75 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VAV00039; U1111-1308-3615 (Other: WHO UTN)
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: RSV Infection; hMPV
Keywords: RSV; RSV Infection; RSV Vaccine; hMPV; hMPV Infection; hMPV Vaccine
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Modified double-blinded for the sentinel and main cohorts.
  * Blinding for vaccine group assignment: participants, outcome assessors, Investigators, laboratory personnel (for both sentinel and main cohort); Sponsor study staff (except biostatistician) and Sponsor SMT (Safety Management Team) for main cohort
  * No blinding for vaccine group assignment: those preparing and administering the study interventions; Sponsor study staff and Sponsor SMT for sentinel cohorts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- Group 1 RSV/hMPV dose A1 (Experimental): Participants will receive a single IM (Intramuscular) injection on day 1 of the RSV/hMPV vaccines according to their randomization schedule.
  Interventions: Biological: RSV/hMPV vaccine dose A1
- Group 2 RSV/hMPV dose A2 (Experimental): Participants will receive a single IM injection on day 1 of the RSV/hMPV vaccines according to their randomization schedule.
  Interventions: Biological: RSV/hMPV vaccine dose A2
- Group 3 RSV/hMPV dose A3 (Experimental): Participants will receive a single IM injection on day 1 of the RSV/hMPV vaccines according to their randomization schedule.
  Interventions: Biological: RSV/hMPV vaccine dose A3
- Group 4 RSV/hMPV dose B1 (Experimental): Participants will receive a single IM injection on day 1 of the RSV/hMPV vaccines according to their randomization schedule.
  Interventions: Biological: RSV/hMPV vaccine dose B1
- Group 5 RSV/hMPV dose B2 (Experimental): Participants will receive a single IM injection on day 1 of the RSV/hMPV vaccines according to their randomization schedule.
  Interventions: Biological: RSV/hMPV vaccine dose B2
- Group 6 RSV/hMPV dose B3 (Experimental): Participants will receive a single IM injection on day 1 of the RSV/hMPV vaccines according to their randomization schedule.
  Interventions: Biological: RSV/hMPV vaccine dose B3
- Group 7 RSV/hMPV dose C1 (Experimental): Participants will receive a single IM injection on day 1 of the RSV/hMPV vaccines according to their randomization schedule.
  Interventions: Biological: RSV/hMPV vaccine dose C1
- Group 8 RSV/hMPV dose C2 (Experimental): Participants will receive a single IM injection on day 1 of the RSV/hMPV vaccines according to their randomization schedule.
  Interventions: Biological: RSV/hMPV vaccine dose C2
- Group 9 RSV/hMPV dose C3 (Experimental): Participants will receive a single IM injection on day 1 of the RSV/hMPV vaccines according to their randomization schedule.
  Interventions: Biological: RSV/hMPV vaccine dose C3
- Group 10 RSV/hMPV dose 1 (Experimental): Participants will receive a single IM injection on day 1 of the RSV/hMPV vaccines according to their randomization schedule.
  Interventions: Biological: RSV/hMPV vaccine dose 1
- Group 11 RSV/hMPV dose 2 (Experimental): Participants will receive a single IM injection on day 1 of the RSV/hMPV vaccines according to their randomization schedule.
  Interventions: Biological: RSV/hMPV vaccine dose 2
- Group 12 RSV/hMPV dose 3 (Experimental): Participants will receive a single IM injection on day 1 of the RSV/hMPV vaccines according to their randomization schedule.
  Interventions: Biological: RSV/hMPV vaccine dose 3
- Group 13 Monovalent RSV Vaccine (Experimental): Participants will receive a single IM injection on day 1 of a Monovalent (MV) RSV vaccine according to their randomization schedule.
  Interventions: Biological: Monovalent RSV Vaccine

INTERVENTIONS:
Biological: RSV/hMPV vaccine dose A1 — Suspension for injection. Route of administration: IM injection
  Arms: Group 1 RSV/hMPV dose A1
Biological: RSV/hMPV vaccine dose A2 — Suspension for injection. Route of administration: IM injection
  Arms: Group 2 RSV/hMPV dose A2
Biological: RSV/hMPV vaccine dose A3 — Suspension for injection. Route of administration: IM injection
  Arms: Group 3 RSV/hMPV dose A3
Biological: RSV/hMPV vaccine dose B1 — Suspension for injection. Route of administration: IM injection
  Arms: Group 4 RSV/hMPV dose B1
Biological: RSV/hMPV vaccine dose B2 — Suspension for injection. Route of administration: IM injection
  Arms: Group 5 RSV/hMPV dose B2
Biological: RSV/hMPV vaccine dose B3 — Suspension for injection. Route of administration: IM injection
  Arms: Group 6 RSV/hMPV dose B3
Biological: RSV/hMPV vaccine dose C1 — Suspension for injection. Route of administration: IM injection
  Arms: Group 7 RSV/hMPV dose C1
Biological: RSV/hMPV vaccine dose C2 — Suspension for injection. Route of administration: IM injection
  Arms: Group 8 RSV/hMPV dose C2
Biological: RSV/hMPV vaccine dose C3 — Suspension for injection. Route of administration: IM injection
  Arms: Group 9 RSV/hMPV dose C3
Biological: RSV/hMPV vaccine dose 1 — Suspension for injection. Route of administration: IM injection
  Arms: Group 10 RSV/hMPV dose 1
Biological: RSV/hMPV vaccine dose 2 — Suspension for injection. Route of administration: IM injection
  Arms: Group 11 RSV/hMPV dose 2
Biological: RSV/hMPV vaccine dose 3 — Suspension for injection. Route of administration: IM injection
  Arms: Group 12 RSV/hMPV dose 3
Biological: Monovalent RSV Vaccine — Suspension for injection. Route of administration: IM injection
  Arms: Group 13 Monovalent RSV Vaccine

SUMMARY:
VAV00039 is a first-in-human (FiH) study to assess the safety and immunogenicity (in adult participants aged 60-75 years) after a single injection of different dose formulations of an RSV/hMPV vaccine candidate and RSV vaccine.

DETAILED DESCRIPTION:
The duration of participation will be approximately 6 months for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 to 75 years on the day of inclusion
* A female participant is eligible to participate if she is post-menopausal for at least 1 year, or surgically sterile

Exclusion Criteria:

* Any condition which, in the opinion of the Investigator, might interfere with the evaluation of the study objectives.
* The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2025-10-09 (Actual)

PRIMARY OUTCOMES:
Presence of any unsolicited systemic Adverse Events (AEs) reported within 30 minutes after vaccination | On Day 1
Presence of solicited injection site and systemic reactions (ie, pre-listed in the participant's diary and in the eCRF (electronic case report form) occurring through 7 days after vaccination | Day 1 through day 8
Presence of unsolicited AEs reported through 28 days after vaccination | Day 1 through day 29
Presence of SAEs (Serious Adverse Events) and AESIs (Adverse Events of Special Interest) throughout the study (ie, through 6 months after vaccination | SAE: Screening through day 181; AESI: Day 1 through day 181
Presence of out-of-range biological test results (including shift from baseline values) through 7 days after vaccination | Screening through day 8

SECONDARY OUTCOMES:
RSV A and RSV B serum nAb (neutralizing antibodies) titers at pre-vaccination and 28 days post-vaccination in all participants | At day 1 and day 29
hMPV A serum nAb titers at pre-vaccination and 28 days post-vaccination in all participants, except in those receiving the MV RSV vaccine | At day 1 and day 28
RSV A and RSV B nAb titers at pre-vaccination, 28 days, 3 months, and 6 months post-vaccination in all participants | At day 1, day 29, day 91, and day 181
RSV A serum anti-F IgG (immunoglobulin type G) Ab (Antibody) titers at pre-vaccination, 28 days, 3 months, and 6 months post-vaccination in all participants | At day 1, day 29, day 91, and day 181
hMPV A nAb titers at pre-vaccination, 28 days, 3 months, and 6 months post-vaccination in all participants, except in those receiving the MV RSV vaccine | At day 1, day 29, day 91, and day 181
hMPV serum anti-F IgG Ab titers at pre-vaccination, 28 days, 3 months, and 6 months post-vaccination in all participants, except in those receiving the MV RSV vaccine | At day 1, day 29, day 91, and day 181

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (6):
  - Site # 0361004, Botany, New South Wales
  - Site # 031001, Brookvale, New South Wales
  - Site # 0361006, Miranda, New South Wales
  - Site # 0361002, Wollongong, New South Wales
  - Site # 0361003, Herston, Queensland
  - Site # 0361005, South Brisbane, Queensland

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org
Supporting Information: Study Protocol, SAP

REFERENCES:
- See also: Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26178&tenant=MT_SNY_9011